CLINICAL TRIAL: NCT02254252
Title: Nicorandil Versus Nitroglycerin for Symptomatic Relief of Angina in Patients With Slow Coronary Flow Phenomenon Visited in Imam Reza Hospital, Mashhad, Iran
Brief Title: Effects of Nicorandil on Angina Symptoms in Patients With Coronary Slow Flow
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Pouya Nezafati, Dr. Pouya Nezafati, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12604
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Results first posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Slow Coronary Flow; Normal, or Near Normal Coronary Angiography; Stable Angina
Keywords: Slow coronary flow phenomenon; Angina pectoris; chest pain; nicroandil
MeSH Terms: conditions — Angina, Stable; Angina Pectoris; Chest Pain | interventions — Nicorandil; Nitroglycerin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitroglycerin (Active Comparator): sustained-release glyceryl trinitrate (6.4mg tablets, two times a day) + standard treatment (an anti-platelet agent, a beta-blocker, an angiotensin converting enzyme inhibitor, and a 3-hydroxy-3-methyl-glutaryl-CoA reductase inhibitor)
  Interventions: Drug: Nitroglycerin
- Nicorandil (Active Comparator): nicorandil (10mg tablets, two times a day) + standard treatment (an anti-platelet agent, a beta-blocker, an angiotensin converting enzyme inhibitor, and a 3-hydroxy-3-methyl-glutaryl-CoA reductase inhibitor)
  Interventions: Drug: Nicorandil

INTERVENTIONS:
Drug: Nicorandil — nicorandil (10mg tablets, two times a day)
  Arms: Nicorandil
Drug: Nitroglycerin — sustained-release glyceryl trinitrate (6.4mg tablets, two times a day)
  Arms: Nitroglycerin

SUMMARY:
Slow coronary flow is an angiographically diagnosed phenomenon defined as delayed opacification of epicardial arteries in the absence of significant arterial narrowing and blockade. Endothelial dysfunction at the level of microarteries have been proposed as the main pathological mechanism in this regard. Available evidence suggest that standard anti-angina medications (e.g. nitroglycerin) that solely target large coronary trunks might not provide adequate symptomatic relief in patients with slow coronary flow phenomenon. It is hypothesized that anti-angina medications which exert vasodilatory effects in large coronary arteries as well as small dividing branches might be superior to nitroglycerin in amelioration of angina symptoms. The present randomized clinical trial was thus designed and conducted to compare the short-term efficacy of nicorandil (a dual-acting anti-angina medication with effects on both large and small coronary vessels) with nitroglycerin in a group of patients with slow coronary flow presented with frequent angina episodes.

ELIGIBILITY:
Inclusion Criteria:

* on coronary angiographic studies, arterial narrowing did not exceed 50% in any of the three main coronary arteries; (
* a delayed opacification in at least one of the main coronary arteries was documented. Delayed opacification was defines as corrected TIMI frame count > 23 fps

Exclusion Criteria:

* comorbid cardiovascular condition other than mild coronary atherosclerosis and coronary slow flow
* refusal to participate
* discontinuation of treatment
* not returning for the follow up visit

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nitroglycerin | Nicorandil
Started | 27 | 27
Completed | 24 | 25
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nitroglycerin | Nicorandil | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (13.3) | 54.6 (11.1) | 54.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 11 | 14 | 25

OUTCOME MEASURES:

1. Primary Outcome: Angina Episode Frequnecy
Description: One month after treatment, patients were asked to determine the frequency of angina episodes in the preceding week.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: episodes per week
Arm/Group | Nitroglycerin | Nicorandil
Number analyzed (Participants) | 24 | 25
episodes per week | 2.28 (0.15) | 1.68 (0.15)

2. Primary Outcome: Angina Episode Intensity
Description: One month after treatment, patients were asked to determine the average intensity of chest pain in experienced episodes using a Likert-type scale of 0 to 10, where 0 indicated lowest intensity/no pain and 10 indicated the highest possible pain experienced.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nitroglycerin | Nicorandil
Number analyzed (Participants) | 24 | 25
units on a scale | 3.89 (0.30) | 3.03 (0.29)

3. Primary Outcome: Canadian Cardiovascular Society (CCS) Grading of Angina Pectoris
Description: One month after treatment, patients were asked to describe the angina episode and based on their descriptions, the CCS class of chest pain was determined. Based on patient's description of the anginal episodes, angina severity was classified into one of CCS class I (angina only with prolonged demanding physical activity), Class II (Slight limitation, with angina only during vigorous physical activity), Class III (Symptoms with everyday living activities), or class IV (angina at rest).
Time Frame: 1 month
Measure: Number; unit: participants
Arm/Group | Nitroglycerin | Nicorandil
Number analyzed (Participants) | 24 | 25
participants
  CCS Class I | 8 | 19
  CCS Class II | 11 | 4
  CCS Class III | 5 | 2

4. Secondary Outcome: Side-effects
Description: Patients were asked and underwent physical examination regarding the common and uncommon side effects attributed to anti-angina medications
Time Frame: 1 month
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Nitroglycerin | Nicorandil
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 0/24 | 4/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nitroglycerin (N=24) | Nicorandil (N=25)
Gastrointestinal discomfort (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No